CLINICAL TRIAL: NCT04504422
Title: Transcranial Direct Current Stimulation to Improve Dual-task Performance in Idiopathic Parkinson's Disease: A Prospective, Single-center, Double-blind, Explorative Clinical Trial
Brief Title: tDCS for Dual-task Performance in Patients With PD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Han Gil Seo, Associate Professor, Seoul National University Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: PD-tDCS-O
Record Dates: First submitted 2020-08-05; First posted 2020-08-07 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Parkinson Disease
Keywords: Parkinson Disease; transcranial direct current stimulation; dual-task performance
MeSH Terms: conditions — Parkinson Disease | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Primary motor cortex (Experimental): The anodic electrode is positioned in the primary motor cortex (Cz) and the cathode electrode on the right orbital frontal cortex (Fp2). The current increases to 2.0 mA over a period of 30 seconds, maintains 2.0 mA for 19 minutes, and decreases to 0 mA over 30 seconds.
  Interventions: Device: transcranial Direct Current Stimulation (tDCS)
- Left dorsolateral prefrontal cortex (Experimental): The anodic electrode is positioned in the left dorsolateral prefrontal cortex (F3) and the cathode electrode on the right orbital frontal cortex (Fp2). The current increases to 2.0 mA over a period of 30 seconds, maintains 2.0 mA for 19 minutes, and decreases to 0 mA over 30 seconds.
  Interventions: Device: transcranial Direct Current Stimulation (tDCS)
- Ventromedial prefrontal cortex (Experimental): The anodic electrode is positioned in the ventromedial prefrontal cortex (Fpz) and the cathode electrode on the left dorsolateral prefrontal cortex (F4). The current increases to 2.0 mA over a period of 30 seconds, maintains 2.0 mA for 19 minutes, and decreases to 0 mA over 30 seconds.
  Interventions: Device: transcranial Direct Current Stimulation (tDCS)
- Sham stimulation (Sham Comparator): The anodic electrode is positioned in the primary motor cortex (Cz) and the cathode electrode on the right orbital frontal cortex (Fp2). The current increases to 2.0 mA during first 30 seconds, decreases to 0 mA over 30 seconds, and then stops supplying for 19 minutes.
  Interventions: Device: transcranial Direct Current Stimulation (tDCS)

INTERVENTIONS:
Device: transcranial Direct Current Stimulation (tDCS) — tDCS was applied for 20 minutes through two saline-soaked sponge electrodes (diameter 6cm) using the YMS-201B (Ybrain Inc, South Korea).

SUMMARY:
The purpose of this study is to investigate the optimal stimulation location of transcranial direct current stimulation to improve the dual-task performance in patients with Parkinson's disease.

DETAILED DESCRIPTION:
Parkinson's disease (PD) is a disease caused by dopamine deficiency in the striatum resulting from the loss of dopaminergic neuronal cells in the cerebral substantia. It is a progressive neurodegenerative disease characterized by motor symptoms including gait disturbance and balance instability. In the early stages of Parkinson's disease, dysfunction of the sensorimotor area of the basal ganglia typically occurs, leading to habitual control hurdles. Accordingly, cognitive efforts are required to perform habitual tasks such as walking, and the automaticity of walking is reduced. Walking performance in a dual-task condition has been used to assess gait automaticity in patients with Parkinson's disease.

Transcranial direct current stimulation (tDCS) is a non-invasive brain stimulation method that can be used to change cortical activity. Recently, there has been growing attention on tDCS as an adjunct tool for rehabilitation. Several tDCS studies in patients with PD have reported the positive results of tDCS on motor function. However, few studies have reported the therapeutic effect of tDCS on the dual-task performance in PD. In addition, inconsistent results have been reported because tDCS protocol has been applied in various way. Therefore, this study aims to investigate an optimized stimulation site of tDCS that could improve the dual-task performance in patients with PD.

ELIGIBILITY:
Inclusion Criteria:

* Clinically diagnosed as idiopathic Parkinson's disease
* modified Hoehn & Yahr stage 2, 2.5, or 3

Exclusion Criteria:

* History of seizure
* Metallic implants, such as cardiac pacemaker or an artificial cochlea
* Patients with inflammation, burns, or wounds in the stimulation area
* Parkinson's disease dementia; cut-off is < 7 of Korean-Montreal Cognitive Assessment for illiterate patients, < 13 for those educated for 0.5-3 years, < 16 for 4-6 years of education, < 19 for 7-9 years of education, and < 20 for 10 or more years of education.
* Severe dyskinesia or severe on-off phenomenon
* Plan to adjust medication at the time of screening
* Sensory abnormalities of the lower extremities, other neurological or orthopedic disease affecting lower extremities, or severe cardiovascular diseases
* Vestibular disease or paroxysmal vertigo
* Pregnant or lactating patients
* Other comorbidities that make it difficult to participate in this study

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2020-11-05 (Actual); Primary Completion 2024-02-13 (Actual); Study Completion 2024-02-13 (Actual)

PRIMARY OUTCOMES:
Cognitive dual-task interference (%) in Timed-up & go test | Immediately after a 20-minute tDCS session
  Percentage of dual-task interference calculated by the difference between dual-task and single-task performance [Percentage of dual-task interference=(Dual-task performance - Single-task performance)/Single-task performance]
Physical dual-task interference (%) in Timed-up & go test | Immediately after a 20-minute tDCS session
  Percentage of dual-task interference calculated by the difference between dual-task and single-task performance [Percentage of dual-task interference=(Dual-task performance - Single-task performance)/Single-task performance]

SECONDARY OUTCOMES:
Timed-up & go test (sec): single task | Immediately after a 20-minute tDCS session
Timed-up & go test (sec): cognitive dual-task | Immediately after a 20-minute tDCS session
Timed-up & go test (sec): physical dual-task | Immediately after a 20-minute tDCS session
Stroop test | Immediately after a 20-minute tDCS session
Trail making test | Immediately after a 20-minute tDCS session
Digit span test | Immediately after a 20-minute tDCS session

CONTACTS AND LOCATIONS:
Overall Officials: Han Gil Seo, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea